CLINICAL TRIAL: NCT03911739
Title: NIDA CTN Protocol 0080: Medication Treatment for Opioid Use Disorder in Expectant Mothers (MOMs): Infant Neurodevelopmental Outcomes (INO) Sub-study
Brief Title: Medication Treatment for Opioid Use Disorder in Expectant Mothers: Infant Neurodevelopmental Outcomes Sub-study
Acronym: MOMs-INO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: T. John Winhusen, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, T. John Winhusen, PhD, Professor; Vice Chair and Division Director of Addiction Sciences, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0429-3; UG1DA013732 (NIH)
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Opioid-Related Disorders; Drug Addiction; Pregnancy Related; Substance Abuse; Drug Abuse; Neonatal Abstinence Syndrome; Neonatal Opiate Withdrawal Syndrome; Drug Abuse in Pregnancy
Keywords: CTN-0080; clinical trials network; medication assisted treatment; pharmacokinetics
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Neonatal Abstinence Syndrome | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BUP-XR (Experimental): Weekly subcutaneous Buprenorphine Injection (CAM2038) during pregnancy. During the 12-month postpartum phase, participants who are breastfeeding will continue receiving subcutaneous Buprenorphine Injection weekly; participants who are not breastfeeding will receive subcutaneous Buprenorphine Injection monthly.
  The target doses will be 24 mg for the weekly formulation and 96 mg for the monthly formulation, but the actual dose may be lower or higher as determined by the prescribing clinician (e.g., based on craving/withdrawal experienced by the participant, etc.).
  Interventions: Drug: Buprenorphine Injection
- BUP-SL (Active Comparator): Daily sublingual buprenorphine, with or without naloxone, based on site preference, during pregnancy and during the 12-month postpartum phase.
  The target dose will be 16 mg daily, but the actual dose may be lower or higher as determined by the prescribing clinician (e.g., based on craving/withdrawal experienced by the participant, etc.).
  Interventions: Drug: Buprenorphine Sublingual Product

INTERVENTIONS:
Drug: Buprenorphine Injection — Weekly and monthly formulations of injectable, extended-release buprenorphine (BUP-XR).
  Other Names: CAM2038
  Arms: BUP-XR
Drug: Buprenorphine Sublingual Product — Sublingual buprenorphine (BUP-SL), administered daily.
  Other Names: Subutex; Suboxone
  Arms: BUP-SL

SUMMARY:
This is a sub-study of NIDA CTN Protocol 0080: Medication Treatment for Opioid Use Disorder in Expectant Mothers (MOMs; Unique protocol ID: 2019-0429-1). Caretakers of the infants delivered by MOMs participants will be offered the opportunity to enroll in this sub-study, which is designed to evaluate the impact of extended-release buprenorphine (BUP-XR), relative to sublingual buprenorphine (BUP-SL), on infant neurodevelopment. The additional data collected in this sub-study will be combined with data from the main MOMs trial.

ELIGIBILITY:
Inclusion Criteria:

* The participant must be the caretaker of an infant that was delivered as part of the MOMs trial (Unique protocol ID: 2019-0429-1).

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Bayley Scales of Infant Development | 24 months post-partum
  The Bayley Scales of Infant Development is considered the gold standard assessment of early child development and includes cognitive, language, fine motor, and gross motor subscales. Subscale scores each range from 1 - 19, with higher scores indicating higher performance.

SECONDARY OUTCOMES:
Bayley Scales of Infant Development | 12 months post-partum
  The Bayley Scales of Infant Development is considered the gold standard assessment of early child development and includes cognitive, language, fine motor, and gross motor subscales. Subscale scores each range from 1 - 19, with higher scores indicating higher performance.
Child Behavior Checklist | 24 months post-partum
  The Child Behavior Checklist includes items that describe behavioral, emotional, and social problems that characterize preschool children.

CONTACTS AND LOCATIONS:
Overall Officials: T. John Winhusen, PhD, Principal Investigator — University of Cincinnati
Locations (10):
- United States (10):
  - Gateway Community Services, Jacksonville, Florida
  - Massachusetts General Hospital HOPE Clinic, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - CODA, Inc., Portland, Oregon
  - Pregnancy Recovery Center at Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah SUPeRAD Clinic, Salt Lake City, Utah
  - Addiction Recovery Services (ARS), Swedish Medical Center, Seattle, Washington
  - Marshall Health MARC Program, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Data will be transmitted by the study Data and Statistics Center to the designated party for de-identification, posting, storing, and archiving on NIDA's Data Share website. Data Share is an online repository of data from studies funded by the National Institute on Drug Abuse. All de-identified individual participant data is expected to be made available.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Kropp FB, Smid MC, Lofwall MR, Wachman EM, Martin PR, Murphy SM, Wilder CM, Winhusen TJ. Collaborative care programs for pregnant and postpartum individuals with opioid use disorder: Organizational characteristics of sites participating in the NIDA CTN0080 MOMs study. J Subst Use Addict Treat. 2023 Jun;149:209030. doi: 10.1016/j.josat.2023.209030. Epub 2023 Apr 4. PMID 37023858

DOCUMENTS (1):
  • Informed Consent Form (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT03911739/ICF_000.pdf